CLINICAL TRIAL: NCT00813033
Title: Creation and Pilot Evaluation of a Patient Decision Aid as an Adjunct to the Consenting Process for Gastrointestinal Endoscopy in a Pediatric Setting
Brief Title: Use of a Patient Decision Aid for Gastrologic Endoscopy in a Pediatric Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Nancy A. Neilan/ MT (ASCP), CCRC Advanced Clinical Coordinator, Children's Mercy Hospitals and Clinics
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CMH080104.2
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Endoscopy
Keywords: create a patient decision aid for endoscopy; evaluate efficacy of a patient decision aid for endoscopy
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient decision aid (Other)
  Interventions: Other: patient decision aid for endoscopy

INTERVENTIONS:
Other: patient decision aid for endoscopy — patient decision aid will be administered at the point of decision making

SUMMARY:
Parents need understandable information in order to make appropriate choices for their child's health care. This is especially true when making decisions about invasive medical procedures. Parents need to understand what will happen, the risks involved, how these risks will be managed and what other options they have before they can decide what is best for their child. The present proposal involves the creation of a novel patient decision aid about the gastro endoscopy procedure, called a "scope." The purpose of the aid is to provide parents with information so they are able to discuss the options with their child's health care providers.

DETAILED DESCRIPTION:
True informed consent depends on effective, bi-directional communication between parents and their child's healthcare providers. Many things affect the quality of the consenting process including the parents' level of health literacy, English proficiency and cultural perspectives. Our long-term goal is to develop a standardized consenting process that ultimately addresses the needs of the patient and the patient's family so that a truly informed decision can occur. The specific hypothesis is that incorporating the use of a multimedia patient decision aid to assist in the education of patients and their families about an invasive medical procedure (i.e. gastro-endoscopy) will improve knowledge and positively impact the ability of the parent to act on this knowledge when making decisions regarding their child's health care.

ELIGIBILITY:
Inclusion Criteria:

* parents or LARs who are considering a gastro-endoscopy for their child

Exclusion Criteria:

* child has previously undergone an endoscopy
* parent of child has undergone an endoscopy
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Validated survey tools will be used to assess change in the consenting parent's knowledge, expectations of outcomes, clarity of values, decision and decision conflict. | immeadiately after completing patient decision aid

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Neilan, MT, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States